CLINICAL TRIAL: NCT02196311
Title: TREATMENT OF SUPRACONDYLAR FRACTURES IN ADOLESCENTS: CLOSED REDUCTION AND CIRCULAR RING EXTERNAL FIXATION VERSUS OPEN REDUCTION AND INTERNAL FIXATION
Brief Title: Treatment Of Supracondylar Fractures Closed Reduction And Circular Ring External Fixation Versus Open Reduction and Internal Fixation
Status: Withdrawn | Type: Observational
Why Stopped: no patient recruited
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaclyn Hill, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-34336
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Supracondylar Humerus Fractures
Keywords: Supracondylar humerus fractures, external fixation, open reduction, and internal fixation.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Supracondylar humerus fractures: We are looking to compare open reduction internal fixation versus circular external fixation for supracondylar humerus fractures.

SUMMARY:
Patients treated with circular external fixation will have better outcomes (as measured by range of motion (ROM), alignment, outcome surveys) than those treated with open reduction and internal fixation (ORIF).

DETAILED DESCRIPTION:
The purpose of this study is to compare patients who undergo ORIF versus circular external fixation for supracondylar humerus fractures in children ages 12-18. We are asking parental permission to collect information about their child's injury, x-rays, obtain ROM measures, collect input from questionnaires, and review other medical information relating to the injury.

The study is NOT about randomizing subjects to treatment, rather we are asking permission to keep track of the decisions that are made about our population's treatment and how it impacts their recovery.

The eligibility criteria is subject's between 12 and 18 years, if supracondylar/periarticular humerus fracture needed operative fixation, and the fracture is unable to be treated with percutaneous skeletal fixation. Patients will be excluded if they have had a previous elbow injury, Osteogenesis imperfecta or another fragile bone disease, elbow stiffness from another cause, or any pre-existing arm weakness.

The outcome measures all enrolled subjects will complete are the QuickDASH and the Pediatric and Adolescent Outcomes Instruments (PODCI). The QuickDASH is a shortened version of the DASH (Disabilities of the Arm, Shoulder and Hand) Outcome Measure which is intended to measure symptoms and functions in people with musculoskeletal disorders of the upper limb. The QuickDASH is valid and reliable and is used for clinical and research purposes. The PODCI is designed to assess patients overall health, pain and ability to participate in normal daily activities in patients under 19 years of age. We will only distribute both questionnaires to the subjects and we are not collecting parent perception.

ELIGIBILITY:
Inclusion Criteria:

* 12 and 18 years old
* Supracondylar/periarticular humerus fracture needed operative fixation
* Fracture is unable to be treated with percutaneous skeletal fixation.

Exclusion Criteria:

* Any previous elbow injury
* Osteogenesis imperfecta or another fragile bone disease
* Elbow stiffness from another cause
* Any pre-existing arm weakness.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients at Texas Children Hospital will undergo either an open reduction with internal fixation or a closed reduction and circular ring external fixation based on the operating surgeon's preference. We do not plan on randomizing or assigning patients that present to Texas Children's Hospital with a supracondylar humerus fracture. Children that consent to participate will strictly continue their follow-up with the physician that performed the surgery. Post-operative course will be noted, physical exam and x-rays followed and outcome surveys obtained and measured intervals.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM), change is being assessed | Initial post-op (first return visit to clinic after surgery), 6 (+/-) weeks, 3(+/-) months, 6 months, 1 year, and 2 years
  Assessing ROM (elbow flexion/extension) in the initial post-operative period and long-term follow-up is an important outcome measure since it correlated with the ability to perform certain tasks with the arm (e.g. reaching head to shampoo/brush hair, reaching mouth to eat, etc.) The visit time frame as outlined above reflects the visits a child would typically return to clinic after surgery for a supracondylar fracture. Every visit will have a threshold of a few weeks to allow the family to return to clinic. These visits are all after the surgery has been performed. For example, the first or initial visit is the first time the patient will return to the hospital after surgery. At this visit the potential participant will be presented with the study materials and given the opportunity to participate. Should the participant participate the visits in the time frame will occur at the give interval.

SECONDARY OUTCOMES:
Treatments, change is being assessed | Initial post-op, 6 weeks, 3 months, 6 months, 1 year, and 2 years
  Evaluating the various treatments for supracondylar humerus fractures, open reduction internal fixation and circular external fixation. The visit time frame as outlined above reflects the visits a child would typically return to clinic after surgery for a supracondylar fracture. Every visit will have a threshold of a few weeks to allow the family to return to clinic. These visits are all after the surgery has been performed. For example, the first or initial visit is the first time the patient will return to the hospital after surgery. At this visit the potential participant will be presented with the study materials and given the opportunity to participate. Should the participant participate the visits in the time frame will occur at the give interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn F Hill, MD, Principal Investigator — Texas Children's Hospital & Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- See also: Texas Children's Hospital - Orthopedics Department — http://www.texaschildrens.org/Locate/Departments-and-Services/Orthopedics/